CLINICAL TRIAL: NCT01490632
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose-Ranging, Phase 2b Study of Baricitinib in Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: A Phase 2b Study of Baricitinib in Participants With Moderate to Severe Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14455; I4V-MC-JADP (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-12-09; First posted 2011-12-13 (Estimated); Results first posted 2017-07-18 (Actual); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Psoriasis; Skin Diseases; Skin Diseases, Papulosquamous
Keywords: Moderate; Severe; Plaque; Chronic
MeSH Terms: conditions — Psoriasis; Skin Diseases; Skin Diseases, Papulosquamous; Lymphoma, Follicular; Plaque, Amyloid; Bronchiolitis Obliterans Syndrome | interventions — baricitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Part A: Placebo administered orally (PO) once daily (QD) for 12 weeks. Part B: Placebo participants stayed on placebo or re-randomized to baricitinib 8 milligram (mg) or 10 mg PO QD for 12 weeks. Part C: Baricitinib participants re-randomized to 4 mg or placebo PO QD for 16 weeks. Part D: Retreated with Part B efficacious dose.
  Interventions: Drug: Placebo
- Baricitinib 2 mg (Experimental): Part A: Baricitinib administered PO QD for initial 12 weeks. Part B: Depending on participant's response, participant was maintained on current dose, or re-randomized to increased dose PO QD for 12 weeks. Part C: Participants re-randomized to half dose or placebo PO QD for 16 weeks. Part D: Participants retreated with Part B efficacious dose for 52 weeks.
  Interventions: Drug: Baricitinib
- Baricitinib 4 mg (Experimental): Part A: Baricitinib administered PO QD for initial 12 weeks. Part B: Depending on participant's response, participant was maintained on current dose, or re-randomized to increased dose PO QD for 12 weeks. Part C: Participants re-randomized to half dose or placebo PO QD for 16 weeks. Part D: Participants retreated with Part B efficacious dose for 52 weeks.
  Interventions: Drug: Baricitinib
- Baricitinib 8 mg (Experimental): Part A: Baricitinib administered PO QD for initial 12 weeks. Part B: Depending on participant's response, participant was maintained on current dose, or re-randomized to increased dose PO QD for 12 weeks. Part C: Participants re-randomized to half dose or placebo PO QD for 16 weeks. Part D: Participants retreated with Part B efficacious dose for 52 weeks.
  Interventions: Drug: Baricitinib
- Baricitinib 10 mg (Experimental): Part A: Baricitinib administered PO QD for initial 12 weeks. Part B: Depending on participant's response, participant was maintained on current dose, or discontinued from the study for 12 weeks. Part C: Participants re-randomized to 4mg dose or placebo PO QD for 16 weeks. Part D: Participants retreated with Part B efficacious dose for 52 weeks.
  Interventions: Drug: Baricitinib

INTERVENTIONS:
Drug: Placebo — Administered orally
  Arms: Placebo
Drug: Baricitinib — Administered orally
  Other Names: LY3009104; INCB028050
  Arms: Baricitinib 10 mg; Baricitinib 2 mg; Baricitinib 4 mg; Baricitinib 8 mg

SUMMARY:
This is a dose-ranging study designed to investigate the efficacy and safety of Baricitinib in the treatment of participants with moderate to severe, chronic plaque psoriasis as assessed by the Psoriasis Area and Severity Index (PASI) score and routine safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* You must have active chronic plaque psoriasis for at least 6 months prior to entry into the study
* You are a candidate for systemic therapy and/or phototherapy
* You must have active plaque psoriasis covering at least 12% body surface area
* You must have Psoriasis Area and Severity Index (PASI) score of at least 12
* You must have Static Physician's Global Assessment (sPGA) score of at least 3

Exclusion Criteria:

* You must not have received a biologic agent/monoclonal antibody within 8 weeks prior to entry into the study
* You must not have prior treatment with an oral Janus kinase (JAK) inhibitor
* You must not have received a systemic psoriasis (Ps) therapy within 4 weeks prior to entry into the study
* You must not have received a phototherapy within 4 weeks prior to entry into the study
* You must not have received a topical Ps therapy with psoralens within 4 weeks prior to entry into the study
* You must not be pregnant or nursing
* If female of childbearing potential or a male, and do not agree to use 2 forms of highly effective methods of birth control for at least 28 days following the last dose of investigational product
* You must not have had symptomatic herpes zoster or herpes simplex infection within 12 weeks or have a history of disseminated/complicated herpes zoster
* You must not have evidence of active infection, such as fever ≥38.0ºC (100.4ºF)
* You must not have a history of active hepatitis B, hepatitis C, or human immunodeficiency virus (HIV)
* You must not be immunocompromised and, in the opinion of the investigator, are at an unacceptable risk for participating in the study
* You must not have known history hypogammaglobulinemia
* You must not have had a serious systemic or local infection within 12 weeks prior to entry into the study
* You must not have been exposed to a live vaccine within 12 weeks prior to entry into the study, or expected to need/receive a live vaccine (including herpes zoster vaccination) during the course of the study
* You must not have had household contact with a person with active tuberculosis (TB) and did not receive appropriate and documented prophylaxis for TB
* You must not have a serious and/or unstable illness that, in the opinion of the investigator, poses an unacceptable risk for the your participation in the study
* You must not have or have had a history of lymphoproliferative disease; or signs or symptoms suggestive of possible lymphoproliferative disease, including lymphadenopathy or splenomegaly; or active primary or recurrent malignant disease; or been in remission from clinically significant malignancy for less than 5 years
* You must not have a history of chronic alcohol abuse or intravenous (IV) drug abuse within the last 2 years
* You must not have donated blood of more than 500 mL within 4 weeks
* You must not have received a topical Ps treatment within 2 weeks prior to entry into the study

  * Exceptions:
  * class 6 (mild, such as desonide) or class 7 (least potent, such as hydrocortisone) topical steroids used on the face, axilla, palms, soles, and/or genitalia
  * non-medicated shampoos (for example, that do not contain corticosteroids, coal tar, or vitamin D3 analogues)
  * emollients that do not contain alpha or beta hydroxyl acids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2011-12; Primary Completion 2012-12 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (35):
- United States (18):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bakersfield, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Santa Monica, California
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miami, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Miramar, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ocala, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alpharetta, Georgia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Arlington Heights, Illinois
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Louisville, Kentucky
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., East Windsor, New Jersey
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Albuquerque, New Mexico
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rochester, New York
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Winston-Salem, North Carolina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Exton, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Philadelphia, Pennsylvania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Austin, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Dallas, Texas
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Salt Lake City, Utah
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Seattle, Washington
- Canada (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kelowna, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Surrey, British Columbia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Peterborough, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Richmond Hill, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Waterloo, Ontario
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sherbrooke, Quebec
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Québec
- Japan (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chiba
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fukuoka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ishikawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kanagawa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Osaka
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Saitama
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tochigi
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toyama
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carolina, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant Psoriasis Area and Severity Index (PASI) score at the conclusion of Part A stratified participants as either Responder (PASI ≥75), Partial Responder (PASI 50 - PASI 74), or Non-Responder (PASI <50).
Pre-assignment Details: Part A: Initial Treatment Period (Weeks 0 up to 12) Part B: Extension or Step-Up Period (Week 12 up to Week 24) Part C: Washout or Step-Down Period (Week 24 up to Week 40) Part D: (Re-Treatment Period up to 52 Weeks)
Groups:
- Part A: Placebo: Placebo administered orally (PO) once daily (QD) for initial 12 weeks. At Week 12, depending on participant's response, dose could be increased to baricitinib 8 mg or 10 mg PO QD for an additional 12 weeks.
- Part A: Baricitinib 2 mg: Baricitinib 2 milligram (mg) administered PO QD for initial 12 weeks. At Week 12, depending on participant's response, dose could be increased to baricitinib 8 mg or 10 mg PO QD for an additional 12 weeks.
- Part A: Baricitinib 4 mg: Baricitinib 4 mg administered PO QD for initial 12 weeks. At Week 12, depending on participant's response, dose could be increased to baricitinib 8 mg or 10 mg PO QD for an additional 12 weeks.
- Part A: Baricitinib 8 mg: Baricitinib 8 mg administered PO QD for initial 12 weeks. At Week 12, depending on participant's response, dose could be increased to baricitinib 10 mg PO QD for an additional 12 weeks.
- Part A: Baricitinib 10 mg: Baricitinib 10 mg administered PO QD for initial 12 weeks. At Week 12, participants who did not achieve at least a PASI 50 were discontinued from the study.
- Part B: Responder - Low Dose: Baricitinib administered 2 mg or 4 mg PO QD maintained at baricitinib 2 mg or 4 mg PO QD, respectively.
- Part B: Responder - High Dose: Baricitinib administered 8 mg or 10 mg PO QD maintained at baricitinib 8 mg or 10 mg PO QD, respectively.
- Part B: Partial- and Non-responder - Placebo to High Dose: Placebo administered PO QD re-randomized to baricitinib 8 mg or 10 mg PO QD.
- Part B: Partial-responder - Low Dose to Low Dose: Baricitinib administered 2 mg or 4mg PO QD. Randomized to remain on the same dose.
- Part B: Partial- and Non-responder - Low Dose to High Dose: Baricitinib administered 2 mg or 4 mg PO QD re-randomized to baricitinib 8 mg or 10 mg PO QD.
- Part B: Partial- and Non-responder - High Dose to High Dose: Baricitinib administered 8 mg or 10 mg PO QD.
- Part B: Placebo Extension: Placebo PO QD maintained on placebo PO QD.
- Part C: Responder - Low Dose to Placebo: Baricitinib 2 mg or 4 mg PO QD re-randomized to placebo PO QD.
- Part C: Responder - Low Dose to ½ Low Dose: Baricitinib administered 2 mg or 4 mg PO QD re-randomized to baricitinib 1 mg or 2 mg PO QD.
- Part C: Responder - High Dose to Placebo: Baricitinib administered 8 mg or 10 mg PO QD re-randomized to placebo PO QD.
- Part C: Responder - High Dose to Low Dose: Baricitinib administered 8 mg PO QD re-randomized to baricitinib 4 mg PO QD. Baricitinib administered 10 mg PO QD re-randomized to baricitinib 4 mg PO QD.
- Part D: Baricitinib 2 mg - Retreatment: Baricitinib 2 mg administrated PO QD (retreatment with Part B efficacious dose) for 52 weeks.
- Part D: Baricitinib 4 mg - Retreatment: Baricitinib 4 mg administrated PO QD (retreatment with Part B efficacious dose) for 52 weeks.
- Part D: Baricitinib 8 mg - Retreatment: Baricitinib 8 mg administrated PO QD (retreatment with Part B efficacious dose) for 52 weeks.
- Part D: Baricitinib 10 mg - Retreatment: Baricitinib 10 mg administrated PO QD (retreatment with Part B efficacious dose) for 52 weeks.
Period: Part A: Initial Treatment Period
Arm/Group | Part A: Placebo | Part A: Baricitinib 2 mg | Part A: Baricitinib 4 mg | Part A: Baricitinib 8 mg | Part A: Baricitinib 10 mg | Part B: Responder - Low Dose | Part B: Responder - High Dose | Part B: Partial- and Non-responder - Placebo to High Dose | Part B: Partial-responder - Low Dose to Low Dose | Part B: Partial- and Non-responder - Low Dose to High Dose | Part B: Partial- and Non-responder - High Dose to High Dose | Part B: Placebo Extension | Part C: Responder - Low Dose to Placebo | Part C: Responder - Low Dose to ½ Low Dose | Part C: Responder - High Dose to Placebo | Part C: Responder - High Dose to Low Dose | Part D: Baricitinib 2 mg - Retreatment | Part D: Baricitinib 4 mg - Retreatment | Part D: Baricitinib 8 mg - Retreatment | Part D: Baricitinib 10 mg - Retreatment
Started | 34 | 32 | 72 | 64 | 69 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Received at Least One Dose of Study Drug | 34 | 32 | 72 | 64 | 69 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 27 | 28 | 67 | 55 | 52 (Includes participants who completed Part A, but discontinued per protocol using Part A PASI score.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 7 | 4 | 5 | 9 | 17 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 2 | 4 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 3 | 1 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Discontinued at Week 12 per protocol | 0 | 0 | 0 | 0 | 9 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part B: Extension or Step-Up Period
Arm/Group | Part A: Placebo | Part A: Baricitinib 2 mg | Part A: Baricitinib 4 mg | Part A: Baricitinib 8 mg | Part A: Baricitinib 10 mg | Part B: Responder - Low Dose | Part B: Responder - High Dose | Part B: Partial- and Non-responder - Placebo to High Dose | Part B: Partial-responder - Low Dose to Low Dose | Part B: Partial- and Non-responder - Low Dose to High Dose | Part B: Partial- and Non-responder - High Dose to High Dose | Part B: Placebo Extension | Part C: Responder - Low Dose to Placebo | Part C: Responder - Low Dose to ½ Low Dose | Part C: Responder - High Dose to Placebo | Part C: Responder - High Dose to Low Dose | Part D: Baricitinib 2 mg - Retreatment | Part D: Baricitinib 4 mg - Retreatment | Part D: Baricitinib 8 mg - Retreatment | Part D: Baricitinib 10 mg - Retreatment
Started | 0 (See Recruitment Details for explanation of Part B participant assignment.) | 0 (See Recruitment Details for explanation of Part B participant assignment.) | 0 (See Recruitment Details for explanation of Part B participant assignment.) | 0 (See Recruitment Details for explanation of Part B participant assignment.) | 0 (See Recruitment Details for explanation of Part B participant assignment.) | 29 (Part A participants randomized to 2 mg or 4 mg with a PASI ≥75 remained on 2 mg or 4 mg.) | 64 (Part A participants randomized to 8 mg or 10 mg with a PASI ≥75 remained on 8 mg or 10 mg.) | 19 (Placebo participants in Part A with a PASI <75 were re-randomized to 8 mg or 10 mg.) | 16 (Part A participants randomized to 2 mg or 4 mg with a PASI ≥50 to <75 remained on 2 mg or 4 mg.) | 50 (Part A participants randomized to 2 mg or 4 mg with a PASI <50 were re-randomized to 8 mg or 10 mg.) | 43 (Part A 10 mg non-responders were discontinued from the study.) | 8 (Part A participants randomized to Placebo remained on Placebo.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 25 | 51 | 13 | 6 | 25 | 22 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 4 | 13 | 6 | 10 | 25 | 21 | 8 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 2 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Completed Part B and Not Moving to PartC | 0 | 0 | 0 | 0 | 0 | 1 | 6 | 6 | 8 | 19 | 16 | 5 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Part C: Washout or Step-Down Period
Arm/Group | Part A: Placebo | Part A: Baricitinib 2 mg | Part A: Baricitinib 4 mg | Part A: Baricitinib 8 mg | Part A: Baricitinib 10 mg | Part B: Responder - Low Dose | Part B: Responder - High Dose | Part B: Partial- and Non-responder - Placebo to High Dose | Part B: Partial-responder - Low Dose to Low Dose | Part B: Partial- and Non-responder - Low Dose to High Dose | Part B: Partial- and Non-responder - High Dose to High Dose | Part B: Placebo Extension | Part C: Responder - Low Dose to Placebo | Part C: Responder - Low Dose to ½ Low Dose | Part C: Responder - High Dose to Placebo | Part C: Responder - High Dose to Low Dose | Part D: Baricitinib 2 mg - Retreatment | Part D: Baricitinib 4 mg - Retreatment | Part D: Baricitinib 8 mg - Retreatment | Part D: Baricitinib 10 mg - Retreatment
Started | 0 | 0 | 0 | 0 | 0 (One participant completed Part B but discontinued without receiving a Part C treatment assignment.) | 0 (Part A participants randomized to 2 mg or 4 mg with a PASI ≥75 remained on 2 mg or 4 mg.) | 0 (Part A participants randomized to 8 mg or 10 mg with a PASI ≥75 remained on 8 mg or 10 mg.) | 0 (Placebo participants in Part A with a PASI <75 were re-randomized to 8 mg or 10 mg.) | 0 (Part A participants randomized to 2 mg or 4 mg with a PASI ≥50 to <75 remained on 2 mg or 4 mg.) | 0 (Part A participants randomized to 2 mg or 4 mg with a PASI <50 were re-randomized to 8 mg or 10 mg.) | 0 (Part A 10 mg non-responders were discontinued from the study.) | 0 (Part A participants randomized to Placebo remained on Placebo.) | 15 (Responders receiving 2 or 4 mg were re-randomized to receive placebo.) | 16 (Responders receiving 2 or 4 mg were re-randomized to receive half of the dose from Part B.) | 55 (Responders receiving 8 or 10 mg were re-randomized to receive placebo.) | 55 (Responders receiving 8 or 10 mg were re-randomized to receive 4 mg.) | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 10 | 6 | 37 | 18 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 10 | 18 | 37 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Not completed — Did Not Qualify for Part D Per Protocol | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 9 | 14 | 34 | 0 | 0 | 0 | 0
Period: Part D: Re-Treatment Period
Arm/Group | Part A: Placebo | Part A: Baricitinib 2 mg | Part A: Baricitinib 4 mg | Part A: Baricitinib 8 mg | Part A: Baricitinib 10 mg | Part B: Responder - Low Dose | Part B: Responder - High Dose | Part B: Partial- and Non-responder - Placebo to High Dose | Part B: Partial-responder - Low Dose to Low Dose | Part B: Partial- and Non-responder - Low Dose to High Dose | Part B: Partial- and Non-responder - High Dose to High Dose | Part B: Placebo Extension | Part C: Responder - Low Dose to Placebo | Part C: Responder - Low Dose to ½ Low Dose | Part C: Responder - High Dose to Placebo | Part C: Responder - High Dose to Low Dose | Part D: Baricitinib 2 mg - Retreatment | Part D: Baricitinib 4 mg - Retreatment | Part D: Baricitinib 8 mg - Retreatment | Part D: Baricitinib 10 mg - Retreatment
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 (Responders receiving 2 or 4 mg were re-randomized to receive placebo.) | 0 (Responders receiving 2 or 4 mg were re-randomized to receive half of the dose from Part B.) | 0 (Responders receiving 8 or 10 mg were re-randomized to receive placebo.) | 0 (Responders receiving 8 or 10 mg were re-randomized to receive 4 mg.) | 3 (Responders who experienced a relapse or flare proceeded for retreatment with 2 mg.) | 13 (Responders who experienced a relapse or flare proceeded for retreatment with 4 mg.) | 19 (Responders who experienced a relapse or flare proceeded for retreatment with 8 mg.) | 37 (Responders who experienced a relapse or flare proceeded for retreatment with 10 mg.)
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 8 | 12 | 30
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 7 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Part A: Placebo: Placebo administered orally once daily for initial 12 weeks. At Week 12, depending on participant's response, dose could be increased to baricitinib 8 mg or 10 mg PO QD for an additional 12 weeks.
- Part A: Baricitinib 2 mg: Baricitinib 2 milligram administered PO QD for initial 12 weeks. At Week 12, depending on participant's response, dose could be increased to baricitinib 8 mg or 10 mg PO QD for an additional 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Part A: Placebo | Part A: Baricitinib 2 mg | Part A: Baricitinib 4 mg | Part A: Baricitinib 8 mg | Part A: Baricitinib 10 mg | Total
Number analyzed (Participants) | 34 | 32 | 72 | 64 | 69 | 271
Age, Customized [Mean (Standard Deviation); unit: Years] | 46.70 (15.144) | 47.81 (15.165) | 47.21 (11.650) | 47.37 (15.829) | 47.43 (10.425) | 47.31 (13.268)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 11 | 9 | 18 | 18 | 18 | 74
  Male | 23 | 23 | 54 | 46 | 51 | 197
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 11 | 12 | 10 | 43
  Not Hispanic or Latino | 30 | 26 | 61 | 52 | 59 | 228
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 7 | 6 | 12 | 9 | 11 | 45
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 1 | 1 | 4 | 7
  White | 26 | 26 | 58 | 52 | 53 | 215
  More than one race | 0 | 0 | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Japan | 4 | 4 | 9 | 8 | 8 | 33
  North America | 30 | 28 | 63 | 56 | 61 | 238
Duration of Psoriasis (Ps) [Mean (Standard Deviation); unit: Years] | 16.42 (14.297) | 15.00 (9.951) | 19.90 (12.766) | 16.56 (11.948) | 16.60 (10.653) | 17.26 (11.995)
Percent Body Surface Area (BSA) Affected by Psoriasis [Mean (Standard Deviation); unit: Percent of BSA] | 23.18 (11.890) | 30.78 (20.523) | 28.61 (18.797) | 28.23 (15.726) | 24.45 (12.079) | 27.04 (16.101)
Baseline Psoriasis Area and Severity Index (PASI) Score [Mean (Standard Deviation); unit: Units on a Scale] — The PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation, erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no psoriasis to 72 for the most severe disease.
  Units on a Scale | 19.06 (6.805) | 21.36 (11.056) | 20.58 (9.438) | 20.24 (7.827) | 19.01 (6.177) | 20.00 (8.228)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index Score ≥75% (PASI 75) Improvement (Efficacy of Baricitinib in Participants With Moderate to Severe Plaque Psoriasis. Measure: Psoriasis Area and Severity Index [PASI])
Description: The PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation (scaling), erythema (redness), and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no psoriasis to 72 for the most severe disease.
Time Frame: Week 12
Population: North American (NA) modified intent-to-treat (mITT) population: All NA randomized participants who received at least one dose of study drug. Non-responders and participants who discontinued study drug any time prior to time point of interest, or discontinued from study, were defined as non-responders for the non-responder imputation (NRI) analysis.
Measure: Number; unit: Percent of Participants
Arm/Group | Part A: Placebo | Part A: Baricitinib 2 mg | Part A: Baricitinib 4 mg | Part A: Baricitinib 8 mg | Part A: Baricitinib 10 mg
Number analyzed (Participants) | 30 | 28 | 63 | 56 | 61
Percent of Participants | 16.7 | 28.6 | 28.6 | 42.9 | 54.1

2. Secondary Outcome: Percentage of Participants Achieving a Static Physician Global Assessment (sPGA) of (0, 1) (Efficacy of Baricitinib in Participants With Moderate to Severe Plaque Psoriasis. Measure: Static Physician Global Assessment [sPGA])
Description: The sPGA is a physician's determination of the participant's psoriasis lesions overall at a given time point categorized by descriptions for induration, erythema, and scaling. For the analysis of responses, the participant's psoriasis is assessed as clear (0), minimal (1), mild (2), moderate (3), severe (4), or very severe (5). An sPGA (0,1) response was defined as a post-baseline sPGA score of 0 or 1 with at least a 2-point improvement from baseline in sPGA score.
Time Frame: Week 12
Population: All randomized participants who received at least one dose of study drug. Non-Responders, as well as all participants who discontinue study treatment at any time prior to the time point of interest, were defined as Non-Responders for the NRI analysis.
Measure: Number; unit: Percent of Participants
Arm/Group | Part A: Placebo | Part A: Baricitinib 2 mg | Part A: Baricitinib 4 mg | Part A: Baricitinib 8 mg | Part A: Baricitinib 10 mg
Number analyzed (Participants) | 34 | 32 | 72 | 64 | 69
Percent of Participants | 14.7 | 15.6 | 25.0 | 29.7 | 34.8

3. Secondary Outcome: Percentage of Participants Achieving an sPGA of (0, 1) (Efficacy of Baricitinib in Participants With Moderate to Severe Plaque Psoriasis. Measure: Static Physician Global Assessment [sPGA])
Description: as for outcome 2
Time Frame: Week 24
Population: as for outcome 2
Measure: Number; unit: Percent of Participants
Arm/Group | Part B: Responder - Low Dose | Part B: Responder - High Dose | Part B: Partial- and Non-responder - Placebo to High Dose | Part B: Partial-responder - Low Dose to Low Dose | Part B: Partial- and Non-responder - Low Dose to High Dose | Part B: Partial- and Non-responder - High Dose to High Dose | Part B: Placebo Extension
Number analyzed (Participants) | 29 | 64 | 19 | 16 | 50 | 43 | 8
Percent of Participants | 55.2 | 64.1 | 47.4 | 37.5 | 24.0 | 27.9 | 50.0

4. Secondary Outcome: Percentage of Participants Achieving an sPGA of (0, 1) (Efficacy of Baricitinib in Participants With Moderate to Severe Plaque Psoriasis. Measure: Static Physician Global Assessment [sPGA])
Description: as for outcome 2
Time Frame: Week 92
Population: as for outcome 2
Measure: Number; unit: Percent of Participants
Arm/Group | Part D: Baricitinib 2 mg - Retreatment | Part D: Baricitinib 4 mg - Retreatment | Part D: Baricitinib 8 mg - Retreatment | Part D: Baricitinib 10 mg - Retreatment
Number analyzed (Participants) | 3 | 13 | 19 | 37
Percent of Participants | 33.3 | 23.1 | 21.1 | 27.0

5. Secondary Outcome: Change From Baseline in Part A in Mean Psoriasis Area and Severity Index (PASI) Total Score to Week 12 (Efficacy of Baricitinib in Participants With Moderate to Severe Plaque Psoriasis. Measure: Psoriasis Area and Severity Index [PASI])
Description: The PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation, erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no Ps to 72 for the most severe disease. Least Squares Means (LS Means) were calculated using an analysis of covariance (ANCOVA) model on the last observation carried forward (LOCF) with treatment group as a fixed effect and baseline PASI score as a continuous covariate.
Time Frame: Baseline Part A, Week 12
Population: All randomized participants who received at least one dose of study drug. Missing values were imputed with the last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Part A: Placebo | Part A: Baricitinib 2 mg | Part A: Baricitinib 4 mg | Part A: Baricitinib 8 mg | Part A: Baricitinib 10 mg
Number analyzed (Participants) | 34 | 32 | 72 | 64 | 69
Units on a Scale | 5.14 (1.370) | 9.40 (1.413) | 9.46 (0.941) | 11.52 (0.997) | 13.93 (0.962)

6. Secondary Outcome: Change From Baseline in Part A in Mean Psoriasis Area and Severity Index (PASI) Total Score to Week 24 (Efficacy of Baricitinib in Participants With Moderate to Severe Plaque Psoriasis: Measure: Psoriasis Area and Severity Index [PASI])
Description: The PASI combines assessments of the extent of body-surface involvement in 4 anatomical regions (head, trunk, arms, and legs) and the severity of desquamation, erythema, and plaque induration/infiltration (thickness) in each region, yielding an overall score of 0 for no Ps to 72 for the most severe disease.
Time Frame: Baseline Part A, Week 24
Population: All randomized participants who received at least one dose of study drug and at least 1 post-baseline observation in Part A at or prior to week 24. Missing values were imputed with the last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Part B: Responder - Low Dose | Part B: Responder - High Dose | Part B: Partial- and Non-responder - Placebo to High Dose | Part B: Partial-responder - Low Dose to Low Dose | Part B: Partial- and Non-responder - Low Dose to High Dose | Part B: Partial- and Non-responder - High Dose to High Dose | Part B: Placebo Extension
Number analyzed (Participants) | 29 | 64 | 19 | 16 | 50 | 43 | 8
Units on a Scale | 15.62 (5.480) | 16.69 (7.399) | 12.94 (6.711) | 12.23 (7.510) | 14.55 (10.493) | 13.67 (9.966) | 13.43 (5.599)

7. Secondary Outcome: Change From Baseline in Part D in Mean Psoriasis Area and Severity Index (PASI) Total Score to Week 92 (Efficacy of Baricitinib in Participants With Moderate to Severe Plaque Psoriasis. Measure: Psoriasis Area and Severity Index [PASI])
Description: as for outcome 6
Time Frame: Baseline Part D, Week 92
Population: All randomized participants who received ≥1 dose of study drug and has 1 post-baseline observation at or prior to week 92. Missing values were imputed with the last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Part D: Baricitinib 2 mg - Retreatment | Part D: Baricitinib 4 mg - Retreatment | Part D: Baricitinib 8 mg - Retreatment | Part D: Baricitinib 10 mg - Retreatment
Number analyzed (Participants) | 3 | 13 | 19 | 37
Units on a Scale | 6.33 (2.836) | 3.25 (4.447) | 5.84 (5.544) | 6.98 (6.456)

8. Secondary Outcome: Change From Baseline Part A in Dermatology Life Quality Index (DLQI) Total Score to Week 12
Description: The DLQI is a simple, participant-administered, 10 question, validated, quality-of-life questionnaire that covers 6 domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include "not at all," "a lot," and "very much," with corresponding scores of 1, 2, and 3, respectively, and unanswered ("not relevant") responses scored as "0." Totals range from 0 to 30 (less to more impairment), and a 5 point change from baseline is considered clinically relevant. Least Square (LS) Means in total DLQI score were calculated using Mixed Model Repeated Measures (MMRM) with baseline score as covariate, treatment, pooled center, visit and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline Part A, Week 12
Population: All randomized participants who received ≥1 dose of study drug in Part A and had ≥1 evaluable post-baseline DLQI observation. Missing values were imputed with the last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Part A: Placebo | Part A: Baricitinib 2 mg | Part A: Baricitinib 4 mg | Part A: Baricitinib 8 mg | Part A: Baricitinib 10 mg
Number analyzed (Participants) | 34 | 32 | 72 | 63 | 68
Units on a Scale | -1.7 (0.98) | -3.4 (1.00) | -4.6 (0.67) | -4.0 (0.71) | -5.1 (0.69)

9. Secondary Outcome: Change From Baseline Part A in Dermatology Life Quality Index (DLQI) Total Score to Week 24
Description: The DLQI is a simple, participant-administered, 10 question, validated, quality-of-life questionnaire that covers 6 domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment. Response categories include "not at all," "a lot," and "very much," with corresponding scores of 1, 2, and 3, respectively, and unanswered ("not relevant") responses scored as "0." Totals range from 0 to 30 (less to more impairment), and a 5 point change from baseline is considered clinically relevant.
Time Frame: Baseline Part A, Week 24
Population: All randomized participants who received ≥1 dose of study drug in Part B and had ≥1 evaluable post-baseline DLQI observation. Missing values were imputed with the last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Part B: Responder - Low Dose | Part B: Responder - High Dose | Part B: Partial- and Non-responder - Placebo to High Dose | Part B: Partial-responder - Low Dose to Low Dose | Part B: Partial- and Non-responder - Low Dose to High Dose | Part B: Partial- and Non-responder - High Dose to High Dose | Part B: Placebo Extension
Number analyzed (Participants) | 29 | 64 | 19 | 16 | 50 | 42 | 6
Units on a Scale | -6.9 (7.53) | -7.0 (8.18) | -3.8 (6.27) | -1.5 (5.92) | -7.8 (6.89) | -4.5 (8.99) | -3.5 (11.76)

10. Secondary Outcome: Change From Baseline Part D in Dermatology Life Quality Index (DLQI) Total Score to Week 92
Description: as for outcome 9
Time Frame: Baseline Part D, Week 92
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Part D: Baricitinib 2 mg - Retreatment | Part D: Baricitinib 4 mg - Retreatment | Part D: Baricitinib 8 mg - Retreatment | Part D: Baricitinib 10 mg - Retreatment
Number analyzed (Participants) | 3 | 13 | 18 | 37
Units on a Scale | -3.3 (4.93) | -0.5 (3.62) | -2.1 (7.40) | -5.0 (6.31)

11. Secondary Outcome: Change From Baseline Part A in Itch Numeric Rating Scale (Itch NRS) Score at Week 12
Description: The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching from Ps is indicated by circling the number that best describes the worst level of itching in the past 24 hours. LS Means were calculated using MMRM with baseline score as covariate, treatment, pooled center, visit and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline Part A, Week 12
Population: All randomized participants who received ≥1 dose of study drug in Part A and had ≥1 evaluable post-baseline Itch NRS observation. Missing values were imputed with the last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Part A: Placebo | Part A: Baricitinib 2 mg | Part A: Baricitinib 4 mg | Part A: Baricitinib 8 mg | Part A: Baricitinib 10 mg
Number analyzed (Participants) | 34 | 32 | 72 | 64 | 69
Units on a Scale | -1.1 (0.48) | -2.8 (0.49) | -3.3 (0.33) | -3.8 (0.35) | -4.7 (0.34)

12. Secondary Outcome: Change From Baseline Part A in Itch Numeric Rating Scale (Itch NRS) Score to Week 24
Description: The Itch NRS is a participant-administered, 11-point horizontal scale anchored at 0 and 10, with 0 representing "no itch" and 10 representing "worst itch imaginable." Overall severity of a participant's itching from Ps is indicated by circling the number that best describes the worst level of itching in the past 24 hours.
Time Frame: Baseline Part A, Week 24
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Part B: Responder - Low Dose | Part B: Responder - High Dose | Part B: Partial- and Non-responder - Placebo to High Dose | Part B: Partial-responder - Low Dose to Low Dose | Part B: Partial- and Non-responder - Low Dose to High Dose | Part B: Partial- and Non-responder - High Dose to High Dose | Part B: Placebo Extension
Number analyzed (Participants) | 29 | 64 | 19 | 16 | 49 | 43 | 8
Units on a Scale | -4.7 (3.52) | -5.6 (2.96) | -5.4 (3.83) | -3.4 (3.69) | -4.1 (3.33) | -3.5 (3.03) | -2.5 (4.11)

13. Secondary Outcome: Change From Baseline Part D in Itch Numeric Rating Scale (Itch NRS) Score to Week 92
Description: as for outcome 12
Time Frame: Baseline Part D, Week 92
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Part D: Baricitinib 2 mg - Retreatment | Part D: Baricitinib 4 mg - Retreatment | Part D: Baricitinib 8 mg - Retreatment | Part D: Baricitinib 10 mg - Retreatment
Number analyzed (Participants) | 3 | 13 | 18 | 37
Units on a Scale | -2.3 (0.58) | -2.5 (3.23) | -2.7 (2.91) | -3.1 (3.38)

14. Secondary Outcome: Change From Baseline Part A in Quick Inventory of Depressive Symptomatology-Self Report 16 Items (QIDS-SR16) Total Score at Week 12
Description: The 16-item QIDS-SR16 version is a widely used validated scale designed to assess the severity of depressive symptoms. The participant was asked to rate the severity and frequency of specific symptoms present over the last 7 days. The QIDS-SR16 total scores range from 0 to 27, where higher scores indicate higher severity of symptoms. LS Means were calculated using MMRM with baseline score as covariate, treatment, pooled center, visit and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline Part A, Week 12
Population: All randomized participants who received ≥1 dose of study drug in Part A and had ≥1 evaluable post-baseline QIDS-SR16 observation. Missing values were imputed with the last observation carried forward (LOCF) method.
Measure: Least Squares Mean (Standard Error); unit: Units on a Scale
Arm/Group | Part A: Placebo | Part A: Baricitinib 2 mg | Part A: Baricitinib 4 mg | Part A: Baricitinib 8 mg | Part A: Baricitinib 10 mg
Number analyzed (Participants) | 31 | 30 | 67 | 63 | 64
Units on a Scale | -0.9 (0.57) | -1.0 (0.58) | -1.0 (0.39) | -0.7 (0.40) | -0.9 (0.40)

15. Secondary Outcome: Change From Baseline Part A in Quick Inventory of Depressive Symptomatology-Self Report 16 Items (QIDS-SR16) Total Score to Week 24
Description: The QIDS-SR16 is a 16-item, self-report instrument intended to assess the existence and severity of symptoms of depression as listed in the American Psychiatric Association's Diagnostic and Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) (APA 1994). A participant is asked to consider each statement as it relates to the way they have felt for the past 7 days. There is a 4-point scale for each item ranging from 0 to 3. The 16 items corresponding to 9 depression domains are summed to give a single score ranging from 0 to 27, with higher scores denoting greater symptom severity. The domains assessed by the instrument include: (1) sad mood, (2) concentration, (3) self-criticism, (4) suicidal ideation, (5) interest, (6) energy/fatigue, (7) sleep disturbance (initial, middle, and late insomnia or hypersomnia), (8) decrease/increase in appetite/weight, and (9) psychomotor agitation/retardation.
Time Frame: Baseline Part A, Week 24
Population: All randomized participants who received ≥1 dose of study drug in Part A and had ≥1 evaluable post-baseline QIDS-SR16 observation. As observed values were used.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Part B: Responder - Low Dose | Part B: Responder - High Dose | Part B: Partial- and Non-responder - Placebo to High Dose | Part B: Partial-responder - Low Dose to Low Dose | Part B: Partial- and Non-responder - Low Dose to High Dose | Part B: Partial- and Non-responder - High Dose to High Dose | Part B: Placebo Extension
Number analyzed (Participants) | 26 | 57 | 19 | 14 | 41 | 38 | 5
Units on a Scale | -1.6 (2.48) | -2.6 (3.80) | -1.4 (3.15) | -1.2 (2.67) | -1.6 (2.99) | -2.2 (4.64) | -3.0 (6.16)

16. Secondary Outcome: Change From Baseline Part D in Quick Inventory of Depressive Symptomatology-Self Report 16 Items (QIDS-SR16) Total Score to Week 92
Description: as for outcome 15
Time Frame: Baseline Part D, Week 92
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Part D: Baricitinib 2 mg - Retreatment | Part D: Baricitinib 4 mg - Retreatment | Part D: Baricitinib 8 mg - Retreatment | Part D: Baricitinib 10 mg - Retreatment
Number analyzed (Participants) | 0 | 4 | 8 | 14
Units on a Scale |  | -0.25 (1.708) | -0.13 (3.796) | -0.86 (2.143)

17. Secondary Outcome: Change From Baseline Part A in European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Scores
Description: The EQ-5D-5L is a standardized measure of health status of the participant. One of two portions of the EQ-5D-5L was used in which a self-perceived health score is assessed using a visual analogue scale (VAS) that ranged from 0 to 100 millimeter (mm), where 0 mm indicated the "worst health you can imagine" and 100 mm indicated the "best health you can imagine". This information is used as a quantitative measure of health outcome. LS Means were calculated using MMRM with baseline score as covariate, treatment, pooled center, visit and treatment-by-visit interaction as fixed effects.
Time Frame: Baseline Part A, Week 12
Population: All randomized participants who received ≥1 dose of study drug in Part A and had ≥1 evaluable post-baseline EQ-5D-5L observation. As observed values were used.
Measure: Least Squares Mean (Standard Error); unit: Millimeter (mm)
Arm/Group | Part A: Placebo | Part A: Baricitinib 2 mg | Part A: Baricitinib 4 mg | Part A: Baricitinib 8 mg | Part A: Baricitinib 10 mg
Number analyzed (Participants) | 27 | 29 | 67 | 60 | 62
Millimeter (mm) | 2.9 (2.55) | 5.7 (2.46) | 6.4 (1.62) | 9.5 (1.71) | 7.8 (1.69)

18. Secondary Outcome: Change From Baseline Part A in European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Scores
Description: The EQ-5D-5L is a standardized measure of health status of the participant. One of two portions of the EQ-5D-5L was used in which a self-perceived health score is assessed using a visual analogue scale (VAS) that ranged from 0 to 100 millimeter (mm), where 0 mm indicated the "worst health you can imagine" and 100 mm indicated the "best health you can imagine". This information is used as a quantitative measure of health outcome.
Time Frame: Baseline Part A, Week 24
Population: as for outcome 17
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Part B: Partial- and Non-responder - Placebo to High Dose; Part B: Partial-responder - Low Dose to Low Dose: Baricitinib administered 2 mg or 4mg PO QD. Randomized to remain on the same dose.
Arm/Group | Part B: Responder - Low Dose | Part B: Responder - High Dose | Part B: Partial- and Non-responder - Placebo to High Dose | Part B: Partial-responder - Low Dose to Low Dose | Part B: Partial- and Non-responder - Low Dose to High Dose | Part B: Partial- and Non-responder - High Dose to High Dose | Part B: Placebo Extension
Number analyzed (Participants) | 28 | 58 | 19 | 14 | 42 | 38 | 6
mm | 8.1 (11.41) | 13.2 (22.06) | 9.6 (10.78) | 9.4 (20.95) | 7.5 (14.47) | 10.5 (19.94) | 7.8 (11.92)

19. Secondary Outcome: Change From Baseline Part D in European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L) Scores
Description: as for outcome 18
Time Frame: Baseline Part D, Week 92
Population: All randomized participants who received ≥1 dose of study drug in Part A and had ≥1 evaluable post-baseline EQ-5D-5L observation. Missing values were imputed with the last observation carried forward (LOCF) method.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Part D: Baricitinib 2 mg - Retreatment | Part D: Baricitinib 4 mg - Retreatment | Part D: Baricitinib 8 mg - Retreatment | Part D: Baricitinib 10 mg - Retreatment
Number analyzed (Participants) | 3 | 13 | 18 | 37
mm | 8.67 (10.263) | 4.00 (26.920) | 4.78 (13.571) | 4.19 (19.727)

20. Secondary Outcome: Percentage of Participants Experiencing Rebound Upon Discontinuation of Study Drug in Part C
Description: Rebound was defined as worsening of psoriasis compared to baseline at Week 0 (for example, PASI score >125% of baseline value) or new pustular, erythrodermic, or more inflammatory psoriasis occurring within 3 months of stopping study drug.
Time Frame: Week 40
Population: All randomized participants who received ≥1 dose of study drug in Part A and participated in Part C.
Measure: Number; unit: Percentage of Participants
Arm/Group | Part C: Responder - Low Dose to Placebo | Part C: Responder - Low Dose to ½ Low Dose | Part C: Responder - High Dose to Placebo | Part C: Responder - High Dose to Low Dose
Number analyzed (Participants) | 15 | 16 | 55 | 55
Percentage of Participants | 0 | 0 | 0 | 0

21. Secondary Outcome: Pharmacokinetics (PK): Maximum Concentration at Steady State of Dosing (Cmax,ss) of Baricitinib
Time Frame: Day 1:15 minutes(m) to 30m and 1hour(h) to 3h Postdose; Week 1:Predose; Week 4:Predose; Week 8:Predose; 15m to 30m and 1h to 3h Postdose, Week 12:Predose; Weeks 14 and 20; Week 24:Predose; Week 28; Week 40. If applicable: Weeks 4, 24, and 52 Post-Relapse
Population: All randomized participants who received ≥1 dose of study drug in Part A, had evaluable PK, and participated in Part C. Some participants received 4mg or 8 mg and increased to 8mg or 10 mg, depending on the response at week 12. Those participants are treated as separate participants in each dose group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole (nM)
Groups:
- Baricitinib 2 mg: Baricitinib 2 milligram administered PO QD for initial 12 weeks. At Week 12, depending on participant's response, dose could be increased to baricitinib 8 mg or 10 mg PO QD for an additional 12 weeks.
- Baricitinib 4 mg: Baricitinib 4 mg administered PO QD for initial 12 weeks. At Week 12, depending on participant's response, dose could be increased to baricitinib 8 mg or 10 mg PO QD for an additional 12 weeks.
- Baricitinib 8 mg: Baricitinib 8 mg administered PO QD for initial 12 weeks. At Week 12, depending on participant's response, dose could be increased to baricitinib 10 mg PO QD for an additional 12 weeks
- Baricitinib 10 mg: Baricitinib 10 mg administered PO QD for initial 12 weeks. At Week 12, participants who did not achieve at least a PASI 50 were discontinued from the study.
Arm/Group | Baricitinib 2 mg | Baricitinib 4 mg | Baricitinib 8 mg | Baricitinib 10 mg
Number analyzed (Participants) | 32 | 72 | 73 | 78
nanomole (nM) | 52.4 (24.7) | 106 (25.9) | 222 (24.4) | 260 (22.9)

22. Secondary Outcome: PK: Area Under the Concentration-Time Curve Versus Time During One Dosing Interval at Steady State (AUC τ,ss)
Time Frame: as for outcome 21
Population: All randomized participants who received ≥1 dose of study drug in Part A, had evaluable PK, and participated in Part A, B or C. Some participants received 4mg or 8 mg and increased to 8mg or 10 mg, depending on the response at week 12. Those participants are treated as separate participants in each dose group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomole*hour (nM*h)
Groups:
- Baricitinib 2 mg: Baricitinib 2 milligram (mg) administered PO QD for initial 12 weeks. At Week 12, depending on participant's response, dose could be increased to baricitinib 8 mg or 10 mg PO QD for an additional 12 weeks.
Arm/Group | Baricitinib 2 mg | Baricitinib 4 mg | Baricitinib 8 mg | Baricitinib 10 mg
Number analyzed (Participants) | 32 | 72 | 73 | 78
nanomole*hour (nM*h) | 462 (40.7) | 975 (41.1) | 2030 (43.3) | 2440 (42.2)

ADVERSE EVENTS:
Groups:
- Part B: Placebo: Placebo PO QD maintained on placebo PO QD.
- Part B: Low Dose: All participants in the following groups (as described in the Participant Flow):
  * Responder Low Dose
  * Partial Responder Low Dose to Low Dose groups.
- Part B: High Dose: All participants in the following groups (as described in the Participant Flow):
  * Responder High Dose
  * Partial and Non-responder Placebo to High Dose
  * Partial and Non-responder Low Dose to High Dose
  * Partial and Non-responder High Dose to High Dose
- Part C: Placebo: All placebo participant groups after study drug re-randomized.
- Part C: Baricitinib: All baricitinib participant groups after study drug re-randomized to various doses.
- Part D: All Baricitinib Doses: All participant dosages following baricitinib retreatment with Part B efficacious dose for 52 weeks.
- Follow-up: Always Placebo: Participants in follow-up with exposure to placebo only during the study. No placebo received during follow-up.
- Follow-up: Ever Used Baricitinib: Participants in follow-up with exposure to any dose of baricitinib during study. No baricitinib received during follow-up.
Arm/Group | Part A: Placebo | Part A: Baricitinib 2 mg | Part A: Baricitinib 4 mg | Part A: Baricitinib 8 mg | Part A: Baricitinib 10 mg | Part B: Placebo | Part B: Low Dose | Part B: High Dose | Part C: Placebo | Part C: Baricitinib | Part D: All Baricitinib Doses | Follow-up: Always Placebo | Follow-up: Ever Used Baricitinib
Serious Adverse Events (participants affected / at risk) | 1/34 | 1/32 | 1/72 | 1/64 | 1/69 | 0/8 | 0/45 | 2/176 | 1/70 | 1/71 | 1/72 | 0/8 | 0/185
Other Adverse Events (participants affected / at risk) | 11/34 | 9/32 | 12/72 | 21/64 | 23/69 | 4/8 | 13/45 | 41/176 | 11/70 | 16/71 | 37/72 | 0/8 | 8/185
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A: Placebo (N=34) | Part A: Baricitinib 2 mg (N=32) | Part A: Baricitinib 4 mg (N=72) | Part A: Baricitinib 8 mg (N=64) | Part A: Baricitinib 10 mg (N=69) | Part B: Placebo (N=8) | Part B: Low Dose (N=45) | Part B: High Dose (N=176) | Part C: Placebo (N=70) | Part C: Baricitinib (N=71) | Part D: All Baricitinib Doses (N=72) | Follow-up: Always Placebo (N=8) | Follow-up: Ever Used Baricitinib (N=185)
Arteriosclerosis coronary artery (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/17 (1) | 0 (0) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Part A: Placebo (N=34) | Part A: Baricitinib 2 mg (N=32) | Part A: Baricitinib 4 mg (N=72) | Part A: Baricitinib 8 mg (N=64) | Part A: Baricitinib 10 mg (N=69) | Part B: Placebo (N=8) | Part B: Low Dose (N=45) | Part B: High Dose (N=176) | Part C: Placebo (N=70) | Part C: Baricitinib (N=71) | Part D: All Baricitinib Doses (N=72) | Follow-up: Always Placebo (N=8) | Follow-up: Ever Used Baricitinib (N=185)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 4 (7) | 1 (1) | 2 (2) | 6 (7) | 6 (6) | 0 (0) | 5 (5) | 9 (10) | 3 (4) | 6 (6) | 12 (14) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 5 (5) | 0 (0) | 1 (1) | 7 (10) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 2 (2)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/16 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 5 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 3 (3) | 5 (5) | 1 (1) | 1 (1) | 3 (3) | 7 (7) | 1 (1) | 1 (2) | 1 (2) | 0 (0) | 0 (0)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/13 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/16 (1) | 0 (0) | 0 (0)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/19 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/16 (1) | 0 (0) | 0 (0)
Salpingo-oophorectomy bilateral (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1/16 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days